CLINICAL TRIAL: NCT02375997
Title: Early Palliative Care With Standard Oncology Care Versus Standard Oncology Care Alone in Metastatic Esophageal Squamous Carcinoma (ESCC) and Gastric Cancer
Brief Title: Early Palliative Care in Metastatic Esophageal Squamous Carcinoma (ESCC) and Gastric Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Shen Lin, Professor, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPC-UPGI
Record Dates: First submitted 2014-10-27; First posted 2015-03-03 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-02

CONDITIONS: Metastatic Esophageal Squamous Carcinoma; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard oncology care plus palliative care (Experimental)
  Interventions: Other: Palliative care
- Standard oncology care (No Intervention)

INTERVENTIONS:
Other: Palliative care — Early nutrition intervention and psychological intervention
  Arms: Standard oncology care plus palliative care

SUMMARY:
The majority of patients with newly diagnosed metastatic ESCC and gastric cancer patients experience a number of physical and psychosocial symptoms related to their cancer. Those patients endure the greatest level of distress from their disease relative to other cancer populations in China. Although new drugs have been applied in recent years, the median overall survival time of metastatic ESCC and GC patients are still around 12 months. Therefore, it is essential to maximize their quality of life (QOL) from the time of diagnosis. Multiple studies demonstrate that symptoms such as pain, fatigue, and anorexia are prevalent at diagnosis and worsen over time. As a result, suffering increases throughout the course of the illness. To be most effective, palliative care with intensive symptom management and psychosocial support should begin at the time of diagnosis, not once life-prolonging therapies have failed. And some studies have revealed that early palliative can even prolong the overall survival time in advanced lung cancer. The investigators then initiated a randomized phase III clinical trial with standard oncology care plus early palliative care or not in metastatic esophageal carcinoma and gastric cancer to observe whether the early palliative can improve the QOL and even prolong the overall survival time in those patients

ELIGIBILITY:
Inclusion Criteria:

* Having signed informed consent
* Age ≥18 years old
* Histologically confirmed esophageal squamous carcinoma and gastric adenocarcinoma, metastatic disease.
* Measurable disease according to the RECIST criteria(diameter of the lesion should be more than 10mm by spiral CT or MRI, more than 20mm by common CT, the date of image should be less than 15 days before enrollment)
* Karnofsky performance status ≥80
* Life expectancy of ≥ 3 month
* WBC > 3,000/mm3, absolute neutrophil count ≥1500/mm3, platelet > 100,000/mm3, Hb > 9g/dl(within 14 days before enrollment),ALT and AST < 2.5 times ULN (≤5 times ULN in patients with liver metastases),Bilirubin level < 1.0 times ULN,Serum AKP < 2.5 times ULN,Serum creatinine < 1.5 times ULN
* No sever complication, such as active gastrointestinal bleeding, perforation, jaundice, obstruction, non-cancerous fever > 38℃；
* Normal ECG and heart function
* Fertile patients must use effective contraception
* Good compliance

Exclusion Criteria:

* Previous treatment of palliative chemotherapy
* Only with Brain or bone metastasis
* No measurable lesions, eg. pleural fluid and ascites
* Suffer from severe heart disease or disease with other important organs
* Chronic diarrhea or renal dysfunction
* Pregnancy or lactation period
* Other previous malignancy within 5 year, except non-melanoma skin cancer Chronic diarrhea
* Mentally abnormal or disable cognition,including CNS metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 592 (Estimated)
Dates: Start 2014-10; Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 2 years
  Time from randomization to death

SECONDARY OUTCOMES:
Quality of life | 2 years
  Measure the scores of quality of life form
Overall response rate | 1 year
  complete response rate plus partial response rate
Adverse event | 2 year
  Number of participants with adverse events as a measure of safety and tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Universtiy Cancer Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Lu Z, Fang Y, Liu C, Zhang X, Xin X, He Y, Cao Y, Jiao X, Sun T, Pang Y, Wang Y, Zhou J, Qi C, Gong J, Wang X, Li J, Tang L, Shen L. Early Interdisciplinary Supportive Care in Patients With Previously Untreated Metastatic Esophagogastric Cancer: A Phase III Randomized Controlled Trial. J Clin Oncol. 2021 Mar 1;39(7):748-756. doi: 10.1200/JCO.20.01254. Epub 2021 Jan 8. PMID 33417481